CLINICAL TRIAL: NCT03720730
Title: Sleep and Appetite Measures as Suicidal Risk Factors in a French- Spanish Cohort of Suicidal Patients.
Brief Title: SmartCriseS - Smartphone Survey of Suicidal Risk
Acronym: SmartCriseS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other); Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); INSERM U1061 Neuropsychiatry Montpellier, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UF 9821
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Personal History of a Recent Suicidal Crisis; Suicidal Ideation; Suicidal Behaviour
Keywords: Suicidal crisis; Suicidal behaviour; Prevention; Smartphone application; Ecological momentary assessment; Psychiatry; Follow-up
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study participants (Experimental): Patients with a recent history of suicidal crisis (within the last 7 days) will use a smartphone application to evaluate sleep, appetite and social parameters.
  Interventions: Other: EMA

INTERVENTIONS:
Other: EMA — The mobile application (EMA) combines an explicit data collection with an implicit one.
  For the explicit data collection with Memind application, patients will have to answer specific questionnaires about sleep, appetite and social factors. Some of the questions will be asked on regular basis, at the same time everyday, while others will be asked randomly during the day (between 9 a.m and 9 p.m).
  The implicit data collecting will be carried out using smartphone sensors (application eB2).

SUMMARY:
Sleep and appetite disorders as well as social exclusion, have been linked to the emergence of suicidal ideation (SI) and suicide attempts.This study aims to evaluate the relationship between those factors and suicidal ideation and behaviour. To assess those factors an ecological momentary assessment (EMA) desing will be used.

EMA will be carried out using 2 applications integrated into the smartphone of participants (Android or iOS), one to make an explicit data collection with questions and another one for the implicit collection of data from mobile sensors.

1044 suicide attempters will be included in three sites and followed for 6 months. Participants will be evaluated at inclusion and at the end of follow-up. The hypothesis is that sleep, appetite and social exclusion factors collected with the smartphone application will be linked to the intensity of death wish, suicidal ideations and suicidal attempts.

An auxiliary study will also be led with 300 patients carrying an actimeter for the 30 first days after inclusion. This will help collecting more accurate data on various sleep parameters.

DETAILED DESCRIPTION:
The proposed study will use ecological momentary assessment (EMA) via smartphone applications (apps) and wearable trackers to examine the relationship between suicidality (wish to die, suicidal ideation and suicide attempt) and changes in sleep quality and disturbed appetite. These behavioral markers, if the hypothesis is proven true, could help predict increased suicidal risk in real-time within a vulnerable population across different cultures.

The study aims to: (1) Establish the extent to which quality of sleep is related to suicide ideation and suicide attempts; (2) Establish the extent to which change in appetite is related to suicide ideation and suicide attempts; (3) Determine the emotional impact of the app when suicidality is assessed; (4) Clarify the timeline of the relationship between sleep disturbances and suicidal behavior; (5) Develop personalized algorithms based on EMA protocol and motor activity markers or "signatures" to assess the risk of suicide attempts.

The hypothesis is that variations in sleep quality will correlate with increased wish to die, suicide ideation and suicide attempts. It is expected that a decrease in sleep quality will be a suicide risk marker especially among young individuals.

This prospective cross-national study will use the infrastructure of an existing network (WORECA). Woreca has defined a common protocol of suicide assessment, data sharing and analysis strategy.

1044 suicide attempters will be included and followed for 6 months. Each participant will be assessed using an EMA protocol via two smartphone apps: (1) One app will ask everyday questions following a dynamic protocol to assess quality of sleep, appetite, suicidal ideation and psychopathology; (2) the other app will record activity using smartphone sensors. Additionally, 300 participants (150 in France and 150 in Spain) will have their sleep phases and other physiological changes during sleep monitored with a wearable armband. Study outcomes include wish to live, wish to die, suicidal ideation, and suicide attempt during the follow-up period.

A multi-level logit regression analysis will be used to account for multiple observations per individual, to identify individual-level (sleep, appetite, socio-demographic, clinical data, treatment data) and site-level characteristics associated with death desire, suicidal ideation or suicide attempt (aim 1 and 2). Hazards models will also be used to relate covariate characteristics (sleep, appetite, sociodemographic, clinical data, treatment data) with time to suicide reattempt during the follow-up period (aim 1 and 2). Data mining (machine learning) techniques will be used to examine risk factors, patterns of illness evolution (aim 3 and 4) and patient stratification by level of suicidal risk (aim 5).

Identifying surrogate markers of suicidality related with physiological functions, which carry less or no stigma for the patients and are easier to report, or have a lower reporting threshold is an essential task. These markers would allow to predict in real-time an increase in suicidal risk within a vulnerable population and ultimately help to prevent and even personalize treatment.Suicidal behaviours, including suicidal ideation, are preventable but to be efficient, prevention needs to rely on the identication of specific risk factors.

ELIGIBILITY:
Inclusion Criteria:

* To be at least 18 years old
* To use a smartphone as a personal phone
* To have consulted in the context of a suicidal crisis within the last 7 days
* To be able to understand the nature, purpose and methodoly of the study.
* To be in a minimal treatment phase (according to the clinician's judgment).
* To accept participating to the study and the 6 months follow-up and to have signed the informed consent

Exclusion Criteria:

* Refusal of participation
* Subject protected by law (guardianship)
* Deprived of liberty Subject (by judicial or administrative decision)
* Diagnosis of a current hypomanic, manic or mixed episode, or a diagnosis of schizoaffective disorder or schizophrenia.
* No affiliation to the social safety system
* Exclusion period in relation to another protocol
* 65 years old patients and older with an MMSE score < 24 at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1044 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2026-01-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Occurrence of suicidal event assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months
  Evaluate the occurrence of a suicidal event with the C-SSRS. The questionnaire includes four subscales. The suicidal ideation severity subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each one ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.

SECONDARY OUTCOMES:
Evaluation of insomnia assessed by ecological momentary assessment (EMA) | 6 months
  Evaluate insomnia with the Insomnia Severity Index (ISI) score using EMA questions. The ISI score ranges from 0 to 27 (higher number indicating more severe insomnia).
Evaluation of insomnia assessed by Insomnia Severity Index (ISI) | 6 months
  Evaluate insomnia with the ISI score. The ISI score ranges from 0 to 27 (higher number indicating more severe insomnia).
Evaluation of appetite assessed by ecological momentary assessment (EMA) | 6 months
  Evaluate appetite using the Council of Nutrition Appetite Questionnaire (CNAQ) score with EMA questions. The CNAQ score ranges from 8 to 40 (a score of less than 28 is cause for concern, with lower number indicating greater risk).
Evaluation of sensibility to social exclusion assessed by ecological momentary assessment (EMA) | 6 months
  Evaluate social sensibility with EMA questions based on the Perceived Social Support and Interpersonal Needs Questionnaire
Evaluation of suicidal ideation intensity assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months
  Evaluate suicidal ideation intensity with the C-SSRS. The severity of suicidal ideation subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Evaluation of the intensity of death wish assessed by ecological momentary assessment (EMA) | 6 months
  Evaluate death wish intensity with analogical scales
Evaluation of suicide attempts severity assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) | 6 months
  Evaluate suicide attempts severity with the C-SSRS. The severity of suicidal ideation subscale ranges from 1 to 5 (with higher number indicating more severe ideation). The intensity of ideation subscale includes 5 questions each ranging from 1 to 5 (with higher number indicating more intense ideation). The suicidal behavior subscale includes 4 yes/no questions. The suicidal behavior lethality subscale inquires about the level of actual or potential medical damage.
Evaluation of sleep duration assessed by Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Evaluate sleep duration with one item from the PSQI (hours of night sleep during the past week) using EMA
Evaluation of sleep duration assessed by Pittsburgh Sleep Quality Index (PSQI) | 6 months
  Evaluate sleep duration with the PSQI at the end of follow-up. The PSQI score ranges from 0 to 21 (lower score indicating healthier sleep quality)
Evaluation of physical activity by eB2 | 6 months
  Evaluate physical activity with smartphone sensors (eB2).

OTHER OUTCOMES:
Evaluation of sleep quantity with the actimeter | 1 month
  Evaluate sleep quantity with the actimeter, only for patients included in the auxiliary study
Evaluation of sleep quantity with the sleep diary | 1 month
  Evaluate sleep quantity with the sleep diary (self-report), only for patients included in the auxiliary study
Evaluation of sleep quality with the actimeter | 1 month
  Evaluate sleep quality with the actimeter. Only for patients included in the auxiliary study.
Evaluation of sleep quality with the sleep diary | 1 month
  Evaluate sleep quality with the sleep diary. Only for patients included in the auxiliary study

CONTACTS AND LOCATIONS:
Locations (2):
- CHU Montpellier, Montpellier, France
- Fundacion Jimenez Diaz Hospital, Madrid, Spain

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Berrouiguet S, Barrigon ML, Castroman JL, Courtet P, Artes-Rodriguez A, Baca-Garcia E. Combining mobile-health (mHealth) and artificial intelligence (AI) methods to avoid suicide attempts: the Smartcrises study protocol. BMC Psychiatry. 2019 Sep 7;19(1):277. doi: 10.1186/s12888-019-2260-y. PMID 31493783